CLINICAL TRIAL: NCT03318211
Title: Continuation Versus Discontinuation of Magnesium Sulfate After Delivery in Women With Severe Preeclampsia. A Randomized Controlled Trial
Brief Title: Discontinuation of Magnesium Sulfate After Delivery in Women With Severe Preeclampsia. A Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14
Record Dates: First submitted 2017-10-19; First posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Preeclampsia Severe
Keywords: preeclampsia; Magnisium sulfate
MeSH Terms: conditions — Pre-Eclampsia | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MgSO4 discontinuation (Active Comparator): after delivery , no Extradoses of MgSO4 were given
  Interventions: Drug: Magnesium Sulfate
- MgSO4 continuation (Active Comparator): After delivery , Mg Sop4 was given at a rate of 1 gram /hour for 24 hours after delivery
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — Intravenous ampules of MgSo4 was given to only to control group after delivery
  Other Names: MgSO4

SUMMARY:
All women with severe preeclmapsia were given a loading dose of 4 g magnesium sulfate IV followed by the maintenance dose of 1 g/h infusion till the delivery. After delivery, women who received magnesium sulfate for 8 hours or more were randomly divided into two groups:

Group I ( 50 cases) No magnesium sulfate received postpartum and Group II ( 50 cases)-magnesium sulfate infusion is given for conventional 24 h postpartum at a rate of 1 gm per hour

DETAILED DESCRIPTION:
All women with severe preeclmapsia were given a loading dose of 4 g magnesium sulfate IV followed by the maintenance dose of 1 g/h infusion till the delivery. After delivery, women who received magnesium sulfate for 8 hours or more were randomly divided into two equal groups:

Group I is the study group: No post partum magnesium sulfate doses were given. Group II is the control group where magnesium sulfate infusion is given for conventional 24 h postpartum at a rate of 1 gm per hour

ELIGIBILITY:
Inclusion Criteria:

* women with severe preeclampsia
* Severe features of preeclampsia include any of the following findings: systolic blood pressure of 160 mmHg or higher, or diastolic blood pressure of 110 mmHg or higher on two occasions at least 4 hours apart while the patient is on bed rest (unless antihypertensive therapy is initiated before that time),thrombocytopenia, impaired liver function, progressive renal insufficiency, pulmonary edema or new onset cerebral or visual disturbances

Exclusion Criteria:

- severe preeclampsia with serum creatinine[1.2 mg/dl 2. previous history of eclampsia 3. Associated maternal medical diseases: pre-existing diabetes mellitus, epilepsy, renal disease.

4. Renal insufficiency. 5. anuric or oliguric urinary out-put under 25 mL/hour. 6. contraindication to the use of magnesium sulfate such as known hypersensitivity to the drug 7. Those with evident hemolysis, elevated liver enzymes, and low platelet count (HELLP) syndrome

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2017-10-25 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
occurrence of convulsions | 48 hours after delivery
  occurrence of eclamptic fits postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Professor

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Diaz V, Long Q, Oladapo OT. Alternative magnesium sulphate regimens for women with pre-eclampsia and eclampsia. Cochrane Database Syst Rev. 2023 Oct 10;10(10):CD007388. doi: 10.1002/14651858.CD007388.pub3. PMID 37815037